CLINICAL TRIAL: NCT04471714
Title: Effects of Baclofen on Presynaptic Inhibition in Humans
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study recruitment was halted due to restrictions and we have decided to not pursue it further.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00090588
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-02

CONDITIONS: Spasticity, Muscle; Spinal Cord Injuries
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries | interventions — Baclofen

STUDY DESIGN:
Intervention Model Description: This is a double blinded, cross-over, retrospective cohort design where the size of the H-reflex and motor unit firing rates will be examined before and after oral intake of baclofen or placebo.
Who Masked: Participant, Investigator
Masking Description: Participants and researchers will be blinded. The research technician will be not be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Experimental): Control participants will come in for two visits. In a randomized manor, they will receive baclofen on one visit and a placebo on the other.
  Interventions: Drug: Baclofen
- Spinal Cord Injury (Experimental): Participants with a spinal cord injury will come in for two visits. In a randomized manor, they will receive baclofen on one visit and a placebo on the other.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Participants will come in for two visits. In a randomized manor, they will receive baclofen on one visit and a placebo on the other. During each visit the soleus H-reflex will be measured and conditioned by common peroneal nerve stimulation to assess presynaptic inhibition.
  Other Names: Placebo

SUMMARY:
This study examines the role of the GABA-B receptor in long-lasting presynaptic inhibition of primary afferents in human participants. Participants will come in for two visits, receiving baclofen (a GABA-B receptor agonist) on one visit and a placebo during the other. Electro-physiological measures will be use during both visit to asses presynaptic inhibition.

DETAILED DESCRIPTION:
The ability to execute purposeful movements relies on sensory information coming from the body. This sensory information tells us where are limbs are in relation to the rest of our body (posture sense), how fast they are moving (kinesthetic sense), how forcefully we are making a contraction (muscular sense) and if we are being contacted by external objects, changes in temperature, pain, etc (somatic sense). Without these senses, the investigators could not make well-controlled movements or navigate in our environment safely. Because of the importance of these sensory inputs, the nervous system has designed a highly regulated system to control the amount and quality of sensory inflow entering into both the spinal cord and brain. The investigators wish to re-investigate how sensory pathways from our body controls the inflow of sensory inputs in adults with and without neurological injury. Specifically, the investigators want to test if the long-lasting suppression of sensory inflow by other sensory nerves is regulated by GABA-B receptors. The investigators will test this by giving participants the GABA-B receptor agonist baclofen. Nerve stimulation and muscle responses will be used to understand how sensory transmission is being controlled in the spinal cord and the GABA-B receptors involvement. Results from these studies will provide important fundamental information about how normal sensory inflow is controlled so that the investigators can better understand how it may be altered after injury to the brain and spinal cord. This information will open new avenues of study into the treatment of sensory-related dysfunction such as spasticity and motor incoordination that occurs after central nervous system injury or disease.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18 and 65 years.
* General good health

Exclusion Criteria:

* Contraindications to baclofen such as a known hypersensitivity to baclofen, renal impairment, stroke, epilepsy, pregnancy and lactation.
* Injury to peripheral nerves or muscles. Injury to nerves or muscles will confound the interpretation of the spinal reflex data.
* Participants with spinal cord injury already taking oral baclofen to manage spasticity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
The effects of baclofen (GABA-B) on Presynaptic Inhibition of primary afferents | 1 year
  Our primary objective is to determine how activation of GABA-B receptors control transmission of sensory afferents as measured by the H-reflex.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gorassini, PhD, Principal Investigator — University of Alberta
Locations (1):
- 524 HMRC, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available to other researchers upon that researchers request.
Time Frame: Upon completion of the study (TBD).
Access Criteria: IPD will be provided to researchers who have contacted the primary investigator and requested additional data. All data will be de-identified.